CLINICAL TRIAL: NCT01667718
Title: Levofloxacin-containing Therapy for Helicobacter Pylori Treatment
Brief Title: Bismuth Improves the Efficacy of Levofloxacin-containing Triple Therapy for Helicobacter Pylori Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. HONG LU, Professor of GI Division, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2012011
Record Dates: First submitted 2012-06-05; First posted 2012-08-17 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Functional Dyspepsia; Peptic Ulcer
Keywords: eradication; helicobacter pylori; bismuth
MeSH Terms: conditions — Peptic Ulcer | interventions — Bismuth; Lansoprazole; Proton Pump Inhibitors; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levofloxacin-triple therapy (Active Comparator): Lansoprazole (Proton Pump Inhibitor), Levofloxacin, Amoxicillin
  Interventions: Drug: Lansoprazole; Drug: Levoﬂoxacin; Drug: Amoxicillin
- Levofloxacin-quadruple therapy (Experimental): Lansoprazole (Proton Pump Inhibitor),Bismuth, Levofloxacin, Amoxicillin
  Interventions: Drug: Bismuth; Drug: Lansoprazole; Drug: Levoﬂoxacin; Drug: Amoxicillin

INTERVENTIONS:
Drug: Bismuth — Bismuth 220mg b.i.d for 2 weeks
  Other Names: Bismuth potassium citrate
  Arms: Levofloxacin-quadruple therapy
Drug: Lansoprazole — Lansoprazole 30 mg b.i.d.for 2 weeks
  Other Names: Proton Pump Inhibitor
Drug: Levoﬂoxacin — Levoﬂoxacin 0.5 q.d. for 2 weeks
Drug: Amoxicillin — Amoxicillin 1 g b.i.d. for 2 weeks

SUMMARY:
To examine and compare the efficacy of 2 week Levofloxacin-containing therapies with and without Bismuth for H.pylori treatment.

DETAILED DESCRIPTION:
The success rate of the standard triple therapy for H. pylori infection is decreasing recently.Fluoroquinolone has been proposed to replace clarithromycin as an alternative in the treatment. However prevalence of H.pylori resistance to Levofloxacin has increased rapidly in our area. The purpose of this study is to observe the efficacy of 14 day Levofloxacin triple therapy-based, bismuth-containing quadruple therapy for H.pylori treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients who presented with upper gastrointestinal symptoms and endoscopically proven H.pylori-positive functional dyspepsia and scarred peptic ulcer

Exclusion Criteria:

* patients with peptic ulcer, previous H.pylori eradication therapy, previous gastric surgery, pregnancy, lactation, major systemic diseases, receipt of anti-secretory therapy, antibiotics or bismuth in the preceding 4 weeks, or allergy to any one of the medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
eradication rate of Helicobacter pylori | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, Principal Investigator — Shanghai Jiao-Tong University School of Medicine Renji Hospital
Locations (1):
- Shanghai Jiao-Tong University School of Medicine Renji Hospital, Shanghai, Shanghai Municipality, China